CLINICAL TRIAL: NCT03837561
Title: Phase Ⅲ, Randomized, Double-Blind, Active Controlled, Multi-Center, Clinical Trial to Evaluate the Efficacy and Safety of CUNOX® in Patients With Moderate to Severe Glabellar Lines
Brief Title: The Efficacy and Safety of CUNOX® in Patients With Moderate to Severe Glabellar Lines
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Medy-Tox (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MT01-RU18GBL301
Record Dates: First submitted 2019-02-07; First posted 2019-02-12 (Actual); Last update posted 2020-07-29 (Actual); Status verified 2020-07

CONDITIONS: Glabellar Frown Lines
MeSH Terms: interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cunox (Experimental): Cunox (botulinum toxin type A), 0.1 mL injected into each of 5 sites once.
  Interventions: Drug: Cunox
- Botox (Active Comparator): Botox (botulinum toxin type A), 0.1 mL injected into each of 5 sites once.
  Interventions: Drug: Botox

INTERVENTIONS:
Drug: Cunox — Inject 4 Units (0.1 mL) of reconstituted investigational product or the comparator intramuscularly into each of 5 sites, 2 in each corrugator muscle and 1 in the procerus muscle for a total dose of 20 Units.
  Arms: Cunox
Drug: Botox — Inject 4 Units (0.1 mL) of reconstituted investigational product or the comparator intramuscularly into each of 5 sites, 2 in each corrugator muscle and 1 in the procerus muscle for a total dose of 20 Units.
  Arms: Botox

SUMMARY:
To Confirm the non-inferiority of CUNOX® to BOTOX® in the glabellar line improvement of moderate to severe glabellar lines.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged between 18 and 65
* Subjects attaining ≥ grade 2 (moderate) in the investigator's rating of the severity of glabellar lines at maximum forced frown
* Subjects who voluntarily sign the informed consent

Exclusion Criteria:

* Subjects with allergy or hypersensitivity to the investigational drugs or their components
* Subjects who are participating in other clinical trials or have participated in clinical trials 30 days before screening
* Subjects who are not eligible for this study at the discretion of the investigator

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Actual)
Dates: Start 2018-12-13 (Actual); Primary Completion 2019-03-12 (Actual); Study Completion 2019-06-03 (Actual)

PRIMARY OUTCOMES:
Glabellar line improvement rate at maximum frown confirmed with investigator's live assessment of glabellar line severity | at 4 weeks after the injection.
  An investigator makes a live assessment of subject's glabellar lines at maximum frown on a 4-grade scale (0 (none), 1 (mild), 2 (moderate) and 3 (severe)) 4 weeks after the administration of the investigational drug or the comparator. 0 or 1 point is considered as "improved" and glabellar line improvement rate is calculated.

CONTACTS AND LOCATIONS:
Locations (1):
- Medical Center Capital-Health, Moscow, Russia